CLINICAL TRIAL: NCT01631799
Title: Outcome of Patients After Total Knee Replacement: A Comparison of Femoral Nerve Block and Epidural Anesthesia. A Randomized, Controlled Trial
Brief Title: Outcome of Patients After Total Knee Replacement: A Comparison of Femoral Nerve Block and Epidural Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Thomas Mencke, PD Dr. Thomas Mencke, University of Rostock
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A 40 2008
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Morbidity; Mortality; Complications; Function
Keywords: epidural anesthesia; femoral block; patient control analgesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral Block (Active Comparator): One group received a femoral block for analgesia after surgery. Ropivacain was administered continuously for three days.
  Interventions: Device: Femoral catheter
- Epidural Analgesia (Active Comparator): One group received an epidural analgesia after surgery for three days.
  Interventions: Device: Epidural catheter

INTERVENTIONS:
Device: Femoral catheter — Femoral catheter was inserted at the beginning of surgery. After surgery ropivacaine was administered continuously for three days. In addition, patients received piritramide via patient-controlled analgesia. The amount of ropivacaine was measured.
  Arms: Femoral Block
Device: Epidural catheter — The epidural catheter was inserted at the beiginning of surgery. After surgery ropivacaine was applied continuously for three days. In addition, patients received piritramide via patient controlled analgesia. The amount of ropivacaine was measured.
  Arms: Epidural Analgesia

SUMMARY:
Total knee replacement is very common in Germany. After surgery patients have severe pain in the knee; initiation of the physiotherapy, however, is important in the first three days after surgery. Continuous femoral blockade and continuous (lumbar) epidural analgesia are commonly used after surgery. Both methods are used in Germany. Both methods have advantages and disadvantages. We wanted to answer the question which method of analgesia - after total knee replacement - is better concerning complications and function (after 3 months) ?

ELIGIBILITY:
Inclusion Criteria:

* age 18 -80 years
* ASA I-III
* Surgery: total knee replacement
* informed consent

Exclusion Criteria:

* obesity
* contraindication for epidural anesthesia
* coagulation disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Function | 3 months after surgery
  3 months after surgery the function of the total knee replacement is testd

SECONDARY OUTCOMES:
Mortality | 28 days after surgery
Morbidity | 28 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mencke, PD Dr., Principal Investigator — Dep. of Anesthesia, University of Rostock
Locations (1):
- University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany